CLINICAL TRIAL: NCT02576847
Title: A Phase 3 Open-Label Extension Study to Evaluate the Long-Term Safety of Omiganan Topical Gel in Subjects With Rosacea
Brief Title: Study to Evaluate the Long-term Safety of a Once-Daily Omiganan Topical Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-006
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Omiganan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Omiganan gel applied once daily
  Interventions: Drug: Omiganan

INTERVENTIONS:
Drug: Omiganan — Topical gel

SUMMARY:
This study evaluates the long-term safety of once-daily application of Omiganan topical gel in subjects with severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male and nonpregnant female subjects, 18 years of age or older.
2. A diagnosis of severe papulopustular rosacea using the Investigator Global Assessment grading scale at baseline
3. Subjects with the presence of telangiectasia at Baseline
4. Subjects with the presence of facial erythema associated with their rosacea at Baseline

Exclusion Criteria:

1. Subjects with steroid rosacea or subtype 3 (phymatous rosacea).
2. Subjects with nodular rosacea
3. Standard exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (15):
  - Fremont, California
  - Miami, Florida
  - Miramar, Florida
  - Tampa, Florida
  - Arlington Heights, Illinois
  - Carmel, Indiana
  - Indianapolis, Indiana
  - Plainfield, Indiana
  - Watertown, Massachusetts
  - Albuquerque, New Mexico
  - New York, New York
  - Nashville, Tennessee
  - Dallas, Texas
  - Pflugerville, Texas
  - Webster, Texas
- Australia (2):
  - Sydney, New South Wales
  - Woolloongabba, Queensland
- Canada (3):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Drummondville, Quebec
- France (2):
  - Cannes
  - Nice
- Bergen op Zoom, Netherlands
- New Zealand (2):
  - Hamilton
  - Wellington
- Gothenburg, Sweden
- United Kingdom (2):
  - Lanarkshire
  - Manchester

REFERENCES:
- [Derived] You Y, Liu H, Zhu Y, Zheng H. Rational design of stapled antimicrobial peptides. Amino Acids. 2023 Apr;55(4):421-442. doi: 10.1007/s00726-023-03245-w. Epub 2023 Feb 12. PMID 36781451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 sites in the USA, Canada, Australia/New Zealand, and Europe from October 2015 to July 2017.
Period: Overall Study
Arm/Group | Treatment
Started | 307
Completed | 170
Not Completed | 137
Not completed — Adverse Event | 27
Not completed — Lost to Follow-up | 22
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 78
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Arm/Group | Treatment
Number analyzed (Participants) | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 243
  >=65 years | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205
  Male | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80
  Not Hispanic or Latino | 227
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 286
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  New Zealand | 34
  Canada | 24
  Netherlands | 1
  United States | 187
  United Kingdom | 6
  Australia | 37
  France | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 1 or More Treatment-related Treatment-Emergent Adverse Events
Description: Number of subjects with 1 or more treatment-related Treatment-Emergent Adverse Events
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 307
participants | 48

ADVERSE EVENTS:
Time Frame: 378 Days
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/307
Serious Adverse Events (participants affected / at risk) | 7/307
Other Adverse Events (participants affected / at risk) | 83/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=307)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=307)
Viral upper respiratory tract infection (Infections and infestations) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 9 (14)
Application site pain (General disorders) | 10 (12)
Application site erythema (General disorders) | 8 (8)
Application site dryness (General disorders) | 7 (7)
Rosacea (Skin and subcutaneous tissue disorders) | 21 (28)
Headache (Nervous system disorders) | 16 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02576847/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02576847/SAP_001.pdf